CLINICAL TRIAL: NCT03790124
Title: Effectiveness of a Multimodal Prophylactic Strategy to Treat Post-dural Puncture Headache: A Retrospective Study
Brief Title: Post-dural Puncture Headache: A Retrospective Study
Status: Completed | Type: Observational
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Efrain Riveros Perez, MD, Assistant Professor. Department of Anesthesiology, Augusta University
Other Study IDs: 1218545
Record Dates: First submitted 2018-12-26; First posted 2018-12-31 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Obstetric Anesthesia Problems; Headache; Epidural; Anesthesia, Headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neuraxial techniques are widely used in obstetric practice to provide analgesia and anesthesia. A common complication associated with neuraxial anesthesia is post-dural puncture headache (PDPH), resulting from unintentional or unintended puncture of the dura mater during insertion of an epidural needle. Incidence of PDPH after spinal anesthesia is very low due to the widespread use of non-cutting small diameter spinal needles. Incidence of "wet tap" during epidural injection has been reported to be 1.5%, with 52-85% of these patients developing PDPH.

When an obstetric patient develops PDPH, institution of an effective treatment is necessary. Although PDPH tends to resolve spontaneously over a couple of weeks, it carries the risk of potential complications. PDPH interfere with the ability of the mother to take care of her baby, increases the risk of chronic headache and limits early ambulation, thereby increasing the risk of venous thrombosis and pulmonary embolism. As important as treating PDPH when it occurs is to prevent it when the dura is accidentally punctured during labor epidural placement. Multiple therapeutic strategies have been reported in the medical literature to prevent this outcome. Preventive measures range from conservative strategies to invasive procedures. Bedrest and hydration have been traditionally recommended to try to prevent PDPH when a wet tap occurs; however, no conclusive evidence supports their use. The use of oral and intravenous caffeine is insufficiently supported by clinical evidence. Epidural morphine and intravenous cosyntropin have been successfully used to prevent PDPH. Epidural injection of normal saline reduces the gradient for CSF leak. The use of saline has shown variable results in different studies. Although the results of some studies show insufficient evidence about its effectiveness, administration of epidural saline is a technique relatively devoid of significant adverse effects.

The institutional protocol recommends the combination of a multimodal approach to prevention of PDPH after accidental dural puncture, based on strategies reported in the medical literature. The protocol consists of the immediate administration of 60 cc of epidural normal saline, followed by two preventive measures administered after delivery. After delivery, 1 mg of intravenous cosyntropin and 3 mg of epidural morphine before catheter removal are administered. This study tests the hypothesis that the multimodal prophylactic protocol described above decreases the incidence of PDPH and the need to perform epidural blood patch, compared to other strategies or no prophylactic management.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients who underwent labor epidural and had accidental dural puncture

Exclusion Criteria:

* History of migraines or chronic headaches
* History of neurological deficits

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant patients who underwent labor epidural analgesia and had accidental dural puncture (wet tap)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Number of cases with Postdural puncture headache | 3 days after delivery
  Number of patients who had wet tap during epidural placement who developed postdural puncture headache

SECONDARY OUTCOMES:
Number of cases of epidural patch placement | 3 days after delivery
  Number of patients who had wet tap during epidural placement who developed postdural puncture and required performance of epidural blood patch

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided